CLINICAL TRIAL: NCT00440258
Title: Dopamine Agonist Cabergoline Reduces Hemoconcentration and Ascites in Hyperstimulated Women Undergoing Assisted Reproduction.
Brief Title: Cabergoline Reduces OHSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLC-AP-404-207-1
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Ovarian hyperstimulation syndrome, dopamine agonists, cabergoline, hemoconcentration, ascites, ovarian perfusion, dopamine receptor 2
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome; Ascites | interventions — Cabergoline; High-Energy Shock Waves; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cabergoline
Procedure: MR
Procedure: Ultrasound
Procedure: Blood Analysis

SUMMARY:
The present study was designed to provide clinical confirmation of Cb2's value as a new approach in the prevention of increased vascular permeability and hemoconcentration, both signs of OHSS in humans, and in order to explore its mechanism of action. To this end, a prospective, randomized, placebo-controlled study was designed in which Cb2 was employed in women at risk of OHSS after gonadotropin administration for ART. Simultaneously, ovarian perfusion was assessed in these patients using MR pharmacokinetic modeling.

DETAILED DESCRIPTION:
Patients and Study design This study was performed in 82 oocyte donors between April 2004 and July 2006. The study protocol was approved by our institution's Ethical Committee and all participants signed a written consent form. The protocol for COH has previously been described (23). Only patients at risk of developing OHSS were included. The definition of risk was the development of 20-30 follicles >12 mm in diameter, and retrieval of >20 oocytes. Once the decision to administer hCG was taken, patients were immediately allocated into two groups based on a computer randomization: the study group initially consisted of 41 patients, but 6 of these were discarded after randomization because <20 oocytes were retrieved despite the development of >20 follicles >12 mm. Thus, a remaining total of 35 patients received one 0.5 mg tablet of Cb2 daily for eight days. The control group was also initially composed of 41 women. However, 7 of these did not meet the criteria of number of oocytes retrieved, and 2 donors decided to withdraw themselves from the study. This left a remaining total of 32 women, all of whom completed the study, and who received a placebo tablet daily for 8 days. Women were monitored every 48 hours from the day of hCG (day 0) until day 8.

On day hCG+4, in order to define ascites, and provided that there was a certain degree of fluid in the pouch of Douglas after ovum pick-up, we employed transvaginal ultrasound (TVU) to measure two major perpendicular diameters of fluid pockets in 15 donors who showed no risk of OHSS. We observed 3.5±2.8 cm2 of fluid in the pelvis in normal conditions. Therefore, the existence of ascites was confirmed when a pocket of peritoneal fluid >9 cm2 was observed when the patient was in lithotomy position (with the gynecological table always at 45º from the floor of the room), which is the result of the mean± 2 standard deviations (SD) of the value found in non-OHSS candidates. TVU scans were performed by the same researcher (CA), who was blind to the treatment to which the patient was submitted. A 6.5 MHz vaginal probe (Voluson 730 Pro V, General Electric, Madrid, Spain) was employed for all TVU scans.

To evaluate the biochemical risk of hemoconcentration, we evaluated hemoglobin, hematocrit, and leukocyte count. Moreover, renal (creatinine) and liver [transaminases: aspartate aminotransferase (AST); alanine aminotransferase (ALT)] functions, and electrolytes (Na, K) were analyzed to ascertain the severity of the syndrome.

Since all women undergoing ART experience a certain degree of discomfort and enlarged ovaries (known as mild OHSS), we centered our attention on analyzing the incidence of moderate and severe OHSS, which were identified according to our modified (24) classification of Golan et al (25). Moderate OHSS was confirmed when a patient presented ultrasonographic evidence of ascites, while diagnosis of severe OHSS required clinical evidence of ascites and/or hydrothorax and breathing difficulties, or one of the following criteria: a) increased blood viscosity due to hemoconcentration (hemoglobin ≥15 g/dl, hematocrit ≥45%, or leukocyte count ≥20,000/mm3); b) coagulation abnormality; c) diminished renal perfusion and function (serum creatinine levels >1.2 mg/dl); d)liver dysfunction: defined when transaminases (AST or ALT) were >40 U/ml (24, 25).

Additionally, serum PRL levels were measured and adverse drug reactions recorded. An end-of-study assessment was scheduled 7-10 days after the last dose of Cb2/placebo.

Moreover, in the first 8 patients included in the study, follicular fluid aspirates without obvious blood contamination were collected, pooled and and mRNA extracted to quantify the amount of Dp-r2 in human ovaries, employing two different molecular techniques.

To further objectively analyze changes in vascular permeability and fluid shifts, confirmatory studies were performed on six women in the study group and four controls, employing magnetic resonance (MR) as described below. Dynamic contrast-enhanced MR was performed at three different stages of the study: at baseline, before gonadotropin administration was initiated; just before hCG injection; and on day hCG+5, after oocyte pick-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years old healthy women, with risk of developing OHSS.

Exclusion Criteria:

* No risk of developing OHSS; < 20 oocytes retrieved.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-04; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pellicer, MD, Study Director — IVI VALENCIA